CLINICAL TRIAL: NCT00344682
Title: A Randomized Double-Blind Pilot Study of Memantine Augmentation in Antidepressant Nonresponders or Incomplete Responders
Brief Title: Memantine Augmentation of Antidepressants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAM-MD-34
Record Dates: First submitted 2006-06-22; First posted 2006-06-27 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Depressive Disorder
Keywords: memantine; Namenda; augmentation; add-on; depression; MDD (major depressive disorder); unipolar depression; NMDA; ketamine; uncompetitive NMDA receptor antagonist
MeSH Terms: conditions — Depressive Disorder; Depression; Depressive Disorder, Major | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- memantine (Experimental): memantine (5-20mg a day)
  Interventions: Drug: memantine
- Placebo (Placebo Comparator): placebo (5-20mg a day)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: memantine — memantine 5mg - 20mg PO daily
  Other Names: Namenda
  Arms: memantine
Drug: Placebo — 5mg - 20mg PO daily over 8 weeks
  Arms: Placebo

SUMMARY:
This study is evaluating the efficacy and safety of the drug memantine (trade name NAMENDA) as an augmentation agent for the treatment of depression in people who are not fully responding to antidepressant medications.

DETAILED DESCRIPTION:
- Objective

The objective of this study is to evaluate the efficacy and safety of 20 mg of memantine administered once daily as an augmentation agent for subjects who have been taking antidepressants for at least 1 month but who have experienced an incomplete or absent therapeutic response.

- Background

Memantine is a moderate affinity, uncompetitive N-methyl-D-aspartate (NMDA) receptor antagonist that is approved for the treatment of moderate-to-severe dementia of the Alzheimer's type. It has been commercially available in 23 countries worldwide since 1982.

There are reports in the published literature that suggest NMDA receptors may be involved in the etiology of depressive disorders. The NMDA antagonist ketamine has been shown to have antidepressant effects in a placebo-controlled clinical trial (Berman et al., 2000). Uncompetitive NMDA receptor antagonists, including memantine, have been shown to exhibit antidepressant-like activity in animal models of depression (Moryl et al., 1993, Papp and Moryl 1994). Animal studies also support the possibility that uncompetitive NMDA receptor antagonists may work synergistically in combination with antidepressants in animal models of depression (Rogoz et al., 2001). Some authors have hypothesized a role for NMDA receptors in the therapeutic effects of numerous antidepressants (Skolnick et al., 1996).

- Study Design and Duration

This is a randomized, single site, double-blind, placebo-controlled, parallel-group study in outpatients. The study consists of an 8-week double-blind treatment period. Approximately 25 patients will be randomized to each treatment group (memantine or placebo) for a total of approximately 50 patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 18 and 85 years of age at screening.
* Patients must provide written informed consent prior to study entry.
* Patients must meet DSM-IV-TR (Diagnostic and Statistical Manual IV Text Revision) criteria for Major Depressive Episode of a severity mild, moderate or severe or in partial remission, as confirmed by the MINI.
* Patients must have a HAM-D (17-item) score of 16 or higher.
* Patients must have been on 1 of the following medications for 4 or more weeks at or above the listed dose with no psychiatric medication dose changes for the past 25 days:

  * 20 mg qD of fluoxetine (Once Daily)
  * 50 mg qD of sertraline
  * 20 mg qD of paroxetine
  * 200 mg qD of fluvoxamine
  * 20 mg qD of citalopram
  * 10 mg qD of escitalopram
  * 150 mg qD of venlafaxine or venlafaxine sustained release
  * 300 mg qD of bupropion or bupropion sustained or extended release
  * 15 mg qD of mirtazapine
  * 60 mg qD of duloxetine
* Participants must agree to keep the dose of their existing antidepressant(s) constant throughout the 8-week trial.

Exclusion Criteria:

* Diagnosis of bipolar disorder or schizophrenic or schizoaffective disorder.
* History of alcohol or drug abuse or dependence within 6 months of enrollment.
* Patients who have received ECT (Electroconvulsive Therapy) in the past 3 months.
* History of seizures.
* Moderate dementia (MMSE score of 20 or less).
* Active suicidal ideation: endorsing a 3 (most severe score) on QIDS-SR (Quick Inventory of Depression Symptomatology Self Reports) suicide item OR a score of 2 or higher for the past week on Suicide Scale items 4 or 5 (current suicidal ideation moderate or strong or would avoid taking steps to save life).
* Currently taking a mood stabilizer or antipsychotic (except lithium clearly used as an augmenting agent).
* Patients who, in the opinion of the investigator, might not be suitable for the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina M Deligiannidis, M.D., Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- Center for Psychopharmacologic Research and Treatment (University of Massachusetts Medical School), Worcester, Massachusetts, United States

REFERENCES:
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Moryl E, Danysz W, Quack G. Potential antidepressive properties of amantadine, memantine and bifemelane. Pharmacol Toxicol. 1993 Jun;72(6):394-7. doi: 10.1111/j.1600-0773.1993.tb01351.x. PMID 8361950
- [Background] Oquendo MA, Baca-Garcia E, Kartachov A, Khait V, Campbell CE, Richards M, Sackeim HA, Prudic J, Mann JJ. A computer algorithm for calculating the adequacy of antidepressant treatment in unipolar and bipolar depression. J Clin Psychiatry. 2003 Jul;64(7):825-33. doi: 10.4088/jcp.v64n0714. PMID 12934985
- [Background] Papp M, Moryl E. Antidepressant activity of non-competitive and competitive NMDA receptor antagonists in a chronic mild stress model of depression. Eur J Pharmacol. 1994 Sep 22;263(1-2):1-7. doi: 10.1016/0014-2999(94)90516-9. PMID 7821340
- [Background] Rogoz Z, Skuza G, Kusmider M, Wojcikowski J, Kot M, Daniel WA. Synergistic effect of imipramine and amantadine in the forced swimming test in rats. Behavioral and pharmacokinetic studies. Pol J Pharmacol. 2004 Mar-Apr;56(2):179-85. PMID 15156068
- [Background] Skolnick P, Layer RT, Popik P, Nowak G, Paul IA, Trullas R. Adaptation of N-methyl-D-aspartate (NMDA) receptors following antidepressant treatment: implications for the pharmacotherapy of depression. Pharmacopsychiatry. 1996 Jan;29(1):23-6. doi: 10.1055/s-2007-979537. PMID 8852530
- [Derived] Dean RL, Hurducas C, Hawton K, Spyridi S, Cowen PJ, Hollingsworth S, Marquardt T, Barnes A, Smith R, McShane R, Turner EH, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with unipolar major depressive disorder. Cochrane Database Syst Rev. 2021 Sep 12;9(9):CD011612. doi: 10.1002/14651858.CD011612.pub3. PMID 34510411
- [Derived] Smith EG, Deligiannidis KM, Ulbricht CM, Landolin CS, Patel JK, Rothschild AJ. Antidepressant augmentation using the N-methyl-D-aspartate antagonist memantine: a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2013 Oct;74(10):966-73. doi: 10.4088/JCP.12m08252. PMID 24229746
- See also: Center for Psychopharmacologic Research and Treatment — http://www.umassmed.edu/psychopharm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited through clinician referral and posted and radio advertising with the majority of patients recruited through clinician referral within our single-site, tertiary-care medical center.
Pre-assignment Details: Participants continued on their previously prescribed antidepressant at the same dose throughout the study.
Groups:
- Placebo: Placebo comparator : 5mg - 20mg PO daily over 8 weeks
- Memantine: memantine : memantine 5mg - 20mg PO daily
Period: Overall Study
Arm/Group | Placebo | Memantine
Started | 16 | 15
Completed | 12 | 14
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Memantine | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 13 | 28
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.75 (11.68) | 54.8 (6.17) | 52.28 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Score (MADRS)
Description: Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. Scores 0 to 6 indicate symptoms absent; 7 to 19 indicates mild depression; 30 to 34 defines moderate; 35 to 60 indicates severe depression. Changes in MADRS score was a primary measure.
Time Frame: Baseline & week 8
Population: The primary outcome examines a mean change in MADRS scores at baseline & week 8 through last observation carried forward (LOCF); no values were imputed for missing assessments. The primary data analysis used intent-to-treat measures and computes final study score minus baseline averaged among participants to evaluate treatment group differences.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 16 | 15
units on a scale | -7.25 (11.14) | -7.13 (6.61)

2. Secondary Outcome: Modified Quick Inventory of Depressive Symptoms Self Report Scale (QIDS-SR)
Description: The 16 item Quick Inventory of Depressive Symptomatology (QIDS-SR16) (Rush et al. 2003) is designed to assess the severity of depressive symptoms, with higher scores representing more severe forms of depression. When complete, the QIDS are scored by summing responses to obtain a total score ranging from 0 to 27. Either appetite increase or decrease, but not both, are used to calculate the total score. Weight increase or decrease, but not both, are used to calculate the total score. Scores 0-5 indicate no severity of depression; 6-10 is mild; 11-15 is moderate; 16-20 is severe; 21-27 is very severe levels of depression. Participants were evaluated at baseline and at weeks 1, 2, 3, 4, 6 & 8.
Time Frame: baseline & week 8
Population: The secondary outcome examines a change over in mean QID-SR scores at baseline & week 8 through last observed data carried forward (LOCF); no values were imputed for missing assessments. Data analysis used intent-to-treat measures and computes final study score minus baseline averaged among participants to evaluate treatment group differences.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 16 | 15
units on a scale | -3.69 (5.00) | -6.47 (5.25)

3. Secondary Outcome: Hamilton Anxiety Rating Scale (HARS)
Description: Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Scores > 30 indicate severe anxiety.
Time Frame: baseline & week 8
Population: Secondary outcome examines a change in mean HARS scores observed at baseline & week 8 through last observed data carried forward (LOCF);no values were imputed for missing assessments.Efficacy data analysis used intent-to-treat measures & computes final study score minus baseline averaged among participants to evaluate treatment group differences
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 16 | 15
units on a scale | -4.13 (5.11) | -5.53 (7.29)

4. Secondary Outcome: Montgomery-Asberg Depression Rating Score (MADRS)
Description: Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6 on 10 items. The overall score ranges from 0 to 60. Scores 0 to 6 indicate symptoms absent; 7 to 19 indicates mild depression; 30 to 34 defines moderate; 35 to 60 indicates severe depression. Changes in response rate and remission rate were assessed for secondary measures.
Time Frame: baseline and week 8
Population: Secondary outcome examines a change in response rates,when 50% change from baseline, & remission rates, when MADRS scores of 12 or less were observed.Fischer exact tests assessed efficiency in each treatment group. Intent-to-treat rates at baseline minus week 8 through last observed data carried forward (LOCF) were used;no data values were imputed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 16 | 15
units on a scale | -10.75 (10.46) | -7.13 (6.11)

ADVERSE EVENTS:
Arm/Group | Placebo | Memantine
Serious Adverse Events (participants affected / at risk) | 1/16 | 1/15
Other Adverse Events (participants affected / at risk) | 3/16 | 3/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Memantine (N=15)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Memantine (N=15)
anxiety (Psychiatric disorders) | 3 (3) | 3 (3)
irritability (Psychiatric disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
Early termination due to slow enrollment, leading to small numbers of subjects enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No